CLINICAL TRIAL: NCT01436708
Title: The Association of Pelvic Organ Prolapse Severity and Urinary Symptoms/Sexual Function
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 100034-F
Record Dates: First submitted 2011-09-18; First posted 2011-09-20 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; urinary symptoms; sexual function
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Women with pelvic organ prolapse often accompany with urinary symptoms or sexual dysfunction, and analyzing the association will be helpful to identify the indication of proper management. Therefore, the aim of this study is to identify the above associations.

ELIGIBILITY:
Inclusion Criteria:

* all cases with with pelvic organ prolapse

Exclusion Criteria:

* nil

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all women with pelvic organ prolapse , especially with cystocele, in our outpatient department or the room of urodynamic studies.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan